CLINICAL TRIAL: NCT01317381
Title: ICG- Livertest Versus New Biomarkers as Prognostic Markers in Critically Ill
Brief Title: ICG- Livertest Versus New Biomarkers as Prognostic Markers in Critically Ill ICG- Livertest Versus New Biomarkers as Prognostic Markers in Critically Ill
Acronym: (Greenpep)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Béchir Markus, PI, CIM
Other Study IDs: Version 2.0. 08.12.2
Record Dates: First submitted 2010-08-23; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2010-08

CONDITIONS: Critically Ill Patients
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ICU patients: Admitted patients to the ICU
  Interventions: Procedure: Observational

INTERVENTIONS:
Procedure: Observational — Blood draw

SUMMARY:
ICG- Leberfunktionstest versus "neue" Biomarker als prognostischer Marker bei intensivmedizischen Patienten

ELIGIBILITY:
Inclusion criteria: Gruppe 1:

* Intensiv-Patienten mit Verbrennungen > 10% der Körperoberfläche
* Alter > 18

Gruppe 2:

* Intensivpatienten nach grossen chirurgischen Eingriffen
* Alter > 18

Gruppe 3:

* Polytraumatisierte, intensivpflichtige Patienten
* Alter > 18

Exclusion criteria: • Alter < 18

* Schwangerschaft
* Einschluss in eine andere Studie
* Moribunde Patienten
* Patienten, die kein Deutsch verstehen
* Jodunverträglichkeit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted ICU Patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Study Completion 2011-05

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland